CLINICAL TRIAL: NCT00895674
Title: Patient Characteristics in Advanced Renal Cell Carcinoma and Daily Practice Treatment With Nexavar
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer HealthCare AG
Other Study IDs: 14686; NX0601; PREDICT; 12649; 12650; 12943; 12808; 12807; 12806; 12755; 12731; 12730; 12944; 13094; 13167; 13209; 13210; 13211; 13274; 13277; 13601; 14178; 14242; 13068; 13121; 13095; 13049
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Carcinoma, Renal Cell; Carcinoma, Renal Cell (Advanced)
Keywords: Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Patients with a diagnosis of advanced RCC

SUMMARY:
Renal cell carcinoma accounts for roughly 3 % of all cancer. It is a rather aggressive cancer type, which means that patients who present with an advanced disease have a rather poor prognosis. When this study has been started the standard therapy for patients has been cytokines, which might be accompanied by significant toxicities or might fail the therapeutic goal. In these cases sorafenib can be a feasible therapeutic option. This non-interventional study has been created and is being conducted to collect clinical data on the patients' therapy with sorafenib in an everyday treatment schedule. The main goal of this study focuses on patient characteristics and tumor status in RCC treated with sorafenib as well as the treatment duration and safety of sorafenib under everyday treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced RCC and decision taken by the investigator to prescribe Sorafenib

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of advanced RCC
Sampling Method: Non-Probability Sample
Enrollment: 2840 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Tumor status | After about 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Treatment duration | At end of study after about 12 months
Safety of sorafenib treatment | At every documented visit for about 12 months
Progression-free survival | Calculation at end of study after about 12 months
Status of Metastases | After about 3, 6, 9 and 12 months
Performance status (ECOG) | After about 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Many Locations, Argentina
- Many Locations, Austria
- Many Locations, China
- Many Locations, Colombia
- Many Locations, Czechia
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Indonesia
- Many Locations, Mexico
- Many Locations, Netherlands
- Many Locations, Philippines
- Many Locations, Poland
- Many Locations, Russia
- Many Locations, Slovakia
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Sweden